CLINICAL TRIAL: NCT01896232
Title: A Multicenter, Multiple-dose, Two-arm, Active-controlled, Double-blind, Double-dummy Study to Compare the Therapeutic Efficacy and Safety of Oral Doses of Cinacalcet HCl With Intravenous Doses of AMG 416 in Hemodialysis Subjects With Secondary Hyperparathyroidism
Brief Title: Head-to-Head Study of Etelcalcetide (AMG 416) and Cinacalcet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20120360; 2013-000192-33 (EudraCT Number)
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Secondary Hyperparathyroidism; Chronic Kidney Disease
Keywords: Secondary Hyperparathyroidism, renal, kidney, kidneys, dialysis, hemodialysis, chronic kidney disease, CKD, SHPT
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic | interventions — etelcalcetide hydrochloride; Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cinacalcet (Active Comparator): Participants were randomized to receive oral cinacalcet once daily and placebo intravenous bolus injection at the end of each hemodialysis session, three times per week (TIW) for 26 weeks. The starting dose of cinacalcet was 30 mg daily and could have been titrated at weeks 5, 9, 13, and 17 to target predialysis serum PTH ≤ 300 pg/mL but no lower than 100 pg/mL while maintaining corrected calcium (cCa) ≥ 8.3 mg/dL.
  Interventions: Drug: Cinacalcet; Drug: Intravenous Placebo
- Etelcalcetide (Experimental): Participants were randomized to receive etelcalcetide administered by intravenous bolus injection at the end of each hemodialysis session TIW, and daily oral doses of placebo tablets for 26 weeks. The starting dose of etelcalcetide was 5 mg, and could have been titrated at weeks 5, 9, 13, and 17 to target predialysis serum PTH ≤ 300 pg/mL but no lower than 100 pg/mL while maintaining cCa ≥ 8.3 mg/dL.
  Interventions: Drug: Etelcalcetide; Drug: Oral Placebo

INTERVENTIONS:
Drug: Etelcalcetide — Administered intravenously three times per week. The starting dose was 5 mg, titrated up to 15 mg based on serum PTH and corrected calcium levels.
  Other Names: AMG 416
  Arms: Etelcalcetide
Drug: Cinacalcet — Cinacalcet was administered orally once a day. The starting dose was 30 mg daily, titrated up to 180 mg daily based on serum PTH and corrected calcium levels.
  Other Names: Sensipar®, Mimpara®
  Arms: Cinacalcet
Drug: Oral Placebo — Administered orally once a day.
  Arms: Etelcalcetide
Drug: Intravenous Placebo — Administered intravenously (IV) three times per week.
  Arms: Cinacalcet

SUMMARY:
The purpose of this study is to demonstrate that treatment with etelcalcetide (AMG 416) is not inferior to treatment with cinacalcet for lowering serum parathyroid hormone (PTH) levels by > 30% from baseline among patients with chronic kidney disease (CKD) and secondary hyperparathyroidism (SHPT) who require management with hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects must be receiving adequate thrice weekly maintenance hemodialysis with a dialysate calcium concentration ≥ 2.5 mEq/L for at least 3 months prior to screening laboratory assessments
* Subjects must have SHPT as defined by one central laboratory screening predialysis serum PTH value > 500 pg/mL, measured on separate days within 2 weeks prior to randomization
* Subjects must have one serum cCa value ≥ 8.3 mg/dL obtained before dialysis within 2 weeks of the date of randomization
* Subjects receiving calcium supplements must have no more than a maximum dose change of 50% within 2 weeks before screening laboratory assessments are obtained, and the dose must remain unchanged through randomization

Exclusion Criteria:

* Eligible subjects cannot have received cinacalcet during the 3 months preceding the first screening laboratory assessment
* Other criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2013-08-13 (Actual); Primary Completion 2014-11-12 (Actual); Study Completion 2015-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (162):
- United States (40):
  - Research Site, Azusa, California
  - Research Site, Bakersfield, California
  - Research Site, Chula Vista, California
  - Research Site, Covina, California
  - Research Site, Granada Hills, California
  - Research Site, La Mesa, California
  - Research Site, La Puente, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, San Gabriel, California
  - Research Site, Whittier, California
  - Research Site, Arvada, Colorado
  - Research Site, Aurora, Colorado
  - Research Site, Longmont, Colorado
  - Research Site, Westminster, Colorado
  - Research Site, Orange, Connecticut
  - Research Site, Pembroke Pines, Florida
  - Research Site, Pinecrest, Florida
  - Research Site, Tampa, Florida
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Southgate, Michigan
  - Research Site, Columbus, Mississippi
  - Research Site, Gulfport, Mississippi
  - Research Site, Sewell, New Jersey
  - Research Site, Great Neck, New York
  - Research Site, Mineola, New York
  - Research Site, Ridgewood, New York
  - Research Site, Rosedale, New York
  - Research Site, The Bronx, New York
  - Research Site, Wilmington, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Fairfax, Virginia
  - Research Site, Portsmouth, Virginia
  - Research Site, Madison, Wisconsin
- Austria (3):
  - Research Site, Feldkirch
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (4):
  - Research Site, Genk
  - Research Site, Hasselt
  - Research Site, Kortrijk
  - Research Site, Roeselare
- Canada (5):
  - Research Site, Edmonton, Alberta
  - Research Site, Saint John, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Brampton, Ontario
  - Research Site, Greenfield Park, Quebec
- Czechia (6):
  - Research Site, Nový Jičín
  - Research Site, Prague
  - Research Site, Praha 4 - Nusle
  - Research Site, Slavkov u Brna
  - Research Site, Třinec
  - Research Site, Ústí nad Orlicí
- Denmark (5):
  - Research Site, Aalborg
  - Research Site, Copenhagen
  - Research Site, Fredericia
  - Research Site, Odense
  - Research Site, Roskilde
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- France (7):
  - Research Site, Boulogne-sur-Mer
  - Research Site, Lille
  - Research Site, Nouilly
  - Research Site, Paris
  - Research Site, Saint-Ouen
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Sainte-Foy-lès-Lyon
- Germany (10):
  - Research Site, Aachen
  - Research Site, Coburg
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Magdeburg
  - Research Site, Mettmann
  - Research Site, Minden
  - Research Site, München
  - Research Site, Wiesbaden
  - Research Site, Zwickau
- Greece (7):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Ioannina
  - Research Site, Larissa
  - Research Site, Nikaia, Piraeus
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hungary (8):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Kaposvár
  - Research Site, Kistarcsa
  - Research Site, Pécs
  - Research Site, Székesfehérvár
  - Research Site, Szigetvár
  - Research Site, Zalaegerszeg
- Italy (10):
  - Research Site, Cagliari
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Lecco
  - Research Site, Lucca
  - Research Site, Milan
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Pordenone
  - Research Site, San Giovanni Rotondo FG
- Latvia (2):
  - Research Site, Riga
  - Research Site, Valmiera
- Lithuania (6):
  - Research Site, Alytus
  - Research Site, Kaunas
  - Research Site, Kėdainiai
  - Research Site, Klaipėda
  - Research Site, Šiauliai
  - Research Site, Ukmerge
- New Zealand (3):
  - Research Site, Hamilton
  - Research Site, Papatoetoe, Auckland
  - Research Site, Takapuna, Auckland City
- Poland (8):
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Poznan
  - Research Site, Sieradz
  - Research Site, Wadowice
  - Research Site, Warsaw
  - Research Site, Zabrze
  - Research Site, Żyrardów
- Portugal (9):
  - Research Site, Almada
  - Research Site, Aveiro
  - Research Site, Estoril
  - Research Site, Forte Da Casa
  - Research Site, Guimarães
  - Research Site, Lisbon
  - Research Site, Santo Tirso
  - Research Site, Setúbal
  - Research Site, Vila Franca de Xira
- Russia (5):
  - Research Site, Mitishi
  - Research Site, Moscow
  - Research Site, Petrozavodsk
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Spain (10):
  - Research Site, Córdoba, Andalusia
  - Research Site, Puerto Real, Andalusia
  - Research Site, Galdakao, Basque Country
  - Research Site, Badalona, Catalonia
  - Research Site, Lleida, Catalonia
  - Research Site, Badajoz, Extremadura
  - Research Site, Pamplona, Navarre
  - Research Site, Torrevieja, Valencia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Sweden (3):
  - Research Site, Malmo
  - Research Site, Stockholm
  - Research Site, Trollhättan
- Switzerland (6):
  - Research Site, Aarau
  - Research Site, Bern
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Locarno
  - Research Site, Zurich
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir

REFERENCES:
- [Background] Block GA, Bushinsky DA, Cheng S, Cunningham J, Dehmel B, Drueke TB, Ketteler M, Kewalramani R, Martin KJ, Moe SM, Patel UD, Silver J, Sun Y, Wang H, Chertow GM. Effect of Etelcalcetide vs Cinacalcet on Serum Parathyroid Hormone in Patients Receiving Hemodialysis With Secondary Hyperparathyroidism: A Randomized Clinical Trial. JAMA. 2017 Jan 10;317(2):156-164. doi: 10.1001/jama.2016.19468. PMID 28097356
- [Background] Stollenwerk B, Iannazzo S, Akehurst R, Adena M, Briggs A, Dehmel B, Parfrey P, Belozeroff V. A Decision-Analytic Model to Assess the Cost-Effectiveness of Etelcalcetide vs. Cinacalcet. Pharmacoeconomics. 2018 May;36(5):603-612. doi: 10.1007/s40273-017-0605-2. PMID 29392552
- [Background] Stollenwerk B, Iannazzo S, Cooper K, Belozeroff V. Exploring the potential value of improved care for secondary hyperparathyroidism with a novel calcimimetic therapy. J Med Econ. 2017 Oct;20(10):1110-1115. doi: 10.1080/13696998.2017.1360309. Epub 2017 Aug 14. PMID 28803497
- [Background] Wu B, Melhem M, Subramanian R, Chen P, Jaramilla Sloey B, Fouqueray B, Hock MB, Skiles GL, Chow AT, Lee E. Clinical Pharmacokinetics and Pharmacodynamics of Etelcalcetide, a Novel Calcimimetic for Treatment of Secondary Hyperparathyroidism in Patients With Chronic Kidney Disease on Hemodialysis. J Clin Pharmacol. 2018 Jun;58(6):717-726. doi: 10.1002/jcph.1090. Epub 2018 Mar 13. PMID 29534286
- [Background] Block GA, Chertow GM, Sullivan JT, Deng H, Mather O, Tomlin H, Serenko M. An integrated analysis of safety and tolerability of etelcalcetide in patients receiving hemodialysis with secondary hyperparathyroidism. PLoS One. 2019 Mar 15;14(3):e0213774. doi: 10.1371/journal.pone.0213774. eCollection 2019. PMID 30875390
- [Background] Wolf M, Block GA, Chertow GM, Cooper K, Fouqueray B, Moe SM, Sun Y, Tomlin H, Vervloet M, Oberbauer R. Effects of etelcalcetide on fibroblast growth factor 23 in patients with secondary hyperparathyroidism receiving hemodialysis. Clin Kidney J. 2019 Apr 26;13(1):75-84. doi: 10.1093/ckj/sfz034. eCollection 2020 Feb. PMID 32082556
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 164 centers in Austria, Belgium, Canada, the Czech Republic, Denmark, Estonia, France, Germany, Greece, Hungary, Italy, Latvia, Lithuania, New Zealand, Poland, Portugal, Russia, Spain, Sweden, Switzerland, Turkey, and the United States. Participants were enrolled from 13 August 2013 to 16 May 2014.
Pre-assignment Details: Eligible participants were stratified by screening serum parathyroid hormone (PTH) level (< 900 or ≥ 900 pg/mL) and region (North America or non-North America) and were randomized 1:1 to receive etelcalcetide intravenously (IV) plus oral placebo or oral cinacalcet plus placebo IV.
Period: Overall Study
Arm/Group | Cinacalcet | Etelcalcetide
Started | 343 | 340
Received Treatment | 341 | 338
Completed | 294 | 287
Not Completed | 49 | 53
Not completed — Death | 6 | 10
Not completed — Withdrawal by Subject | 32 | 31
Not completed — Sponsor Decision | 2 | 0
Not completed — Lost to Follow-up | 9 | 12

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS), defined as all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cinacalcet | Etelcalcetide | Total
Number analyzed (Participants) | 343 | 340 | 683
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (14.4) | 54.0 (13.8) | 54.7 (14.1)
Age, Customized [Number; unit: participants]
  < 65 years | 243 | 262 | 505
  ≥ 65 years | 100 | 78 | 178
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 148 | 299
  Male | 192 | 192 | 384
Race [Number; unit: participants]
  Asian | 7 | 9 | 16
  Black | 52 | 54 | 106
  Native Hawaiian or Other Pacific Islander | 3 | 6 | 9
  White | 277 | 261 | 538
  Other | 4 | 10 | 14
Ethnicity [Number; unit: participants]
  Hispanic/Latino | 41 | 38 | 79
  Not Hispanic/Latino | 302 | 302 | 604
Stratification Factor: Screening Serum Parathyroid Hormone (PTH) [Number; unit: participants]
  < 900 pg/mL | 171 | 169 | 340
  ≥ 900 pg/mL | 172 | 171 | 343
Stratification Factor: Region [Number; unit: participants]
  North America | 105 | 103 | 208
  Non-North America | 238 | 237 | 475
Parathyroid Hormone [Mean (Standard Deviation); unit: pg/mL] | 1138.71 (706.77) | 1092.12 (622.81) | 1115.52 (666.22)
Corrected Calcium [Mean (Standard Deviation); unit: mg/dL] | 9.58 (0.67) | 9.67 (0.71) | 9.62 (0.69)
Phosphorus [Mean (Standard Deviation); unit: mg/dL] — Data available for 341 and 337 participants in each treatment group respectively.
  mg/dL | 5.82 (1.58) | 5.81 (1.69) | 5.81 (1.63)
Corrected Calcium Phosphorus Product (cCa x P) [Mean (Standard Deviation); unit: mg²/dL²] — Data available for 341 and 337 participants in each treatment group respectively.
  mg²/dL² | 55.65 (15.37) | 56.36 (17.15) | 56.00 (16.27)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With > 30% Reduction From Baseline in Mean Parathyroid Hormone During the Efficacy Assessment Phase - Non-inferiority Analysis
Time Frame: Baseline and the efficacy assessment phase (EAP; defined as Weeks 20 to 27, inclusive).
Population: Full analysis set participants with PTH data during the EAP
Measure: Number; unit: percentage of participants
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 310 | 298
percentage of participants | 63.9 | 77.9
Statistical Analysis 1: Comparison: Cinacalcet vs Etelcalcetide; The analysis was conducted on the Full Analysis Set (683 participants). Imputation under the non-inferiority null method was applied to participants who did not have PTH data during the EAP. The Mantel-Haenszel estimator was used to calculate the treatment difference between the proportions (Cinacalcet - Etelcalcetide) stratified by screening PTH level and region; Test type: Non-Inferiority or Equivalence — Etelcalcetide was considered non-inferior to cinacalcet if the upper bound of the 2-sided 95% confidence interval (CI) of the treatment difference (cinacalcet - etelcalcetide) was < 12%, the prespecified margin for non-inferiority; Stratified Treatment Difference = -10.48, 95% CI 2-sided [-17.45 to -3.51]

2. Secondary Outcome: Percentage of Participants With > 50% Reduction From Baseline in Mean PTH During the Efficacy Assessment Phase
Time Frame: Baseline and the efficacy assessment phase (Weeks 20 to 27, inclusive).
Population: Full analysis set; participants were considered non-responders if they did not have PTH data during the EAP (ie, non-responder imputation).
Measure: Number; unit: percentage of participants
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 343 | 340
percentage of participants | 40.2 | 52.4
Statistical Analysis 1: Comparison: Cinacalcet vs Etelcalcetide; Achievement of > 50% reduction in mean predialysis serum PTH from baseline during the EAP was analyzed using the Cochran-Mantel-Haenszel (CMH) test stratified by screening PTH level and region. Superiority of etelcalcetide compared with cinacalcet was tested at the 5% significance level (2-sided); Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.21 to 2.23] — The CMH-stratified odds ratio is Etelcalcetide : Cinacalcet

3. Secondary Outcome: Percentage of Participants With > 30% Reduction From Baseline in Mean PTH During the Efficacy Assessment Phase
Time Frame: Baseline and the efficacy assessment phase (Week 20 to Week 27)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 343 | 340
percentage of participants | 57.7 | 68.2
Statistical Analysis 1: Comparison: Cinacalcet vs Etelcalcetide; Achievement of > 30% reduction in mean predialysis serum PTH from baseline during the EAP was analyzed using the Cochran-Mantel-Haenszel test stratified by screening PTH level and region. Superiority of etelcalcetide compared with cinacalcet was tested at the 5% significance level (2-sided); Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.16 to 2.17] — The CMH stratified odds ratio is Etelcalcetide : Cinacalcet

4. Secondary Outcome: Mean Number of Days of Vomiting or Nausea Per Week in the First 8 Weeks
Description: Participants completed the Nausea/Vomiting Symptom Assessment (NVSA) questionnaire daily. This questionnaire asked participants to indicate the severity of nausea on a scale from 0 (no nausea) to 10 (as severe as can be imagined) and if they had vomited in the past 24 hours. A day of vomiting or nausea was defined as those where the severity of nausea score was > 0 or where the episodes of vomiting score was > 0.
Time Frame: First 8 weeks
Population: Full analysis set with available data. For participants providing less than 7 days of responses to NVSA questions in any given week, data from that week did not contribute to the analysis.
Measure: Least Squares Mean (Standard Error); unit: days of vomiting or nausea per week
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 324 | 331
days of vomiting or nausea per week | 0.3 (0.03) | 0.4 (0.04)
Statistical Analysis 1: Comparison: Cinacalcet vs Etelcalcetide; Analyzed using a generalized linear mixed model with Poisson regression, including screening value of the number of days of nausea and vomiting, treatment, stratification factors (screening PTH level and region), study weeks, and treatment by study weeks as covariates. Superiority of etelcalcetide compared with cinacalcet was tested at the 5% significance level (2-sided); Test type: Superiority or Other; p = 0.27, Generalized Linear Mixed Model; Treatment Rate Ratio = 1.2, 95% CI 2-sided [0.89 to 1.49], Standard Error of Mean 0.15 — The treatment rate ratio is Etelcalcetide : Cinacalcet

5. Secondary Outcome: Percent Change From Baseline in Mean Corrected Calcium During the Efficacy Assessment Phase
Time Frame: Baseline and the efficacy assessment phase (weeks 20 - 27)
Population: Full analysis set with available data.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 310 | 298
percent change | -6.28 (0.44) | -9.83 (0.49)
Statistical Analysis 1: Comparison: Cinacalcet vs Etelcalcetide; Analyzed using a repeated measures mixed effects model, including treatment group, randomization stratification factors (screening PTH level and region), study week, and study week by treatment as fixed effects; Test type: Superiority or Other; Treatment difference = -3.48, 95% CI 2-sided [-4.76 to -2.21], Standard Error of Mean 0.65 — Treatment difference is Etelcalcetide - Cinacalcet

6. Secondary Outcome: Percentage of Participants With Mean Predialysis Serum Phosphorus ≤ 4.5 mg/dL During the Efficacy Assessment Phase
Time Frame: Efficacy assessment phase (weeks 20 - 27)
Population: Full analysis set; participants with no phosphorus assessments during the EAP were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 343 | 340
percentage of participants | 29.2 | 32.1
Statistical Analysis 1: Comparison: Cinacalcet vs Etelcalcetide; Analyzed using the Cochran-Mantel-Haenszel method stratified by screening PTH level and region; Test type: Superiority or Other; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.83 to 1.59] — The CMH-stratified odds ratio is Etelcalcetide : Cinacalcet

7. Secondary Outcome: Mean Severity of Nausea in the First 8 Weeks
Description: Severity of nausea was assessed using the Nausea and Vomiting Symptom Assessment questionnaire which asked participants to rate the severity of nausea on a scale from 0 (no nausea) to 10 (as severe as can be imagined). For each participant, the mean severity of nausea was calculated by averaging all available daily severities (including zeroes) reported in the first 8 weeks.
Time Frame: First 8 weeks
Population: Full analysis set with available data
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 339 | 339
units on a scale | 0.48 (0.06) | 0.45 (0.06)
Statistical Analysis 1: Comparison: Cinacalcet vs Etelcalcetide; Analyzed using an analysis of covariance (ANCOVA) model adjusted for screening PTH level and region; Test type: Superiority or Other; Treatment Difference = -0.03, 95% CI 2-sided [-0.18 to 0.12], Standard Error of Mean 0.08 — Treatment difference is Etelcalcetide - Cinacalcet

8. Secondary Outcome: Mean Number of Episodes of Vomiting Per Week in the First 8 Weeks
Description: The number of vomiting episodes was assessed using the Nausea and Vomiting Symptom Assessment questionnaire which asks participants on a daily basis how many times they vomited in the past 24 hours. The number of episodes in a week is the sum of all reported daily episodes in the week.
  For participants providing less than 7 days of responses to NVSA questions in any given week, data from that week did not contribute to the analysis.
Time Frame: First 8 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: vomiting episodes per week
Arm/Group | Cinacalcet | Etelcalcetide
Number analyzed (Participants) | 324 | 331
vomiting episodes per week | 0.1 (0.02) | 0.2 (0.02)
Statistical Analysis 1: Comparison: Cinacalcet vs Etelcalcetide; This analysis was conducted using a generalized linear mixed model with Poisson regression including screening value of the number of episodes of vomiting, treatment, stratification factors (screening PTH level and region), study weeks, and treatment by study weeks as covariates; Test type: Superiority or Other; Treatment Rate Ratio = 1.2, 95% CI 2-sided [0.86 to 1.72], Standard Error of Mean 0.22 — The treatment rate ratio is Etelcalcetide : Cinacalcet

ADVERSE EVENTS:
Time Frame: From Day 1 until 30 days after the last dose; the treatment period was 26 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Cinacalcet | Etelcalcetide
Serious Adverse Events (participants affected / at risk) | 93/341 | 85/338
Other Adverse Events (participants affected / at risk) | 259/341 | 278/338
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cinacalcet (N=341) | Etelcalcetide (N=338)
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 3 | 2
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1
Duodenitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 1
Device malfunction (General disorders) | 0 | 1
Device occlusion (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Medical device complication (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Arteriovenous graft site abscess (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 3 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 2 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 4
Gastroenteritis (Infections and infestations) | 1 | 2
Infected fistula (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pharyngolaryngeal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 1 | 2
Renal cyst infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 4 | 3
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 1 | 0
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 2 | 2
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 1
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 3 | 0
Haemodialysis complication (Injury, poisoning and procedural complications) | 1 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 3 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 3 | 0
Vascular injury (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Blood calcium decreased (Investigations) | 1 | 1
Colonoscopy (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Calciphylaxis (Metabolism and nutrition disorders) | 1 | 1
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Brown tumour (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Altered state of consciousness (Nervous system disorders) | 2 | 0
Amputation stump pain (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Depression suicidal (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Sopor (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Aortic arteriosclerosis (Vascular disorders) | 1 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0
Brachiocephalic vein stenosis (Vascular disorders) | 2 | 0
Extremity necrosis (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 2
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 2
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Venous stenosis (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cinacalcet (N=341) | Etelcalcetide (N=338)
Anaemia (Blood and lymphatic system disorders) | 11 | 17
Diarrhoea (Gastrointestinal disorders) | 34 | 21
Nausea (Gastrointestinal disorders) | 77 | 62
Vomiting (Gastrointestinal disorders) | 46 | 44
Blood calcium decreased (Investigations) | 203 | 232
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 17
Muscle spasms (Musculoskeletal and connective tissue disorders) | 20 | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 17
Headache (Nervous system disorders) | 24 | 21
Hypertension (Vascular disorders) | 22 | 20
Hypotension (Vascular disorders) | 10 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.